CLINICAL TRIAL: NCT04387071
Title: The Seena Magowitz Phase IB/II Trial of CMP-001 (a TLR9 Agonist) in Combination With INCAGN01949 (an Activating Anti-OX40 Antibody) for In Situ Intratumoral Injection for Patients With Stage IV Pancreatic and Other Cancers Except Melanoma
Brief Title: CMP-001 and INCAGN01949 for Patients With Stage IV Pancreatic Cancer and Other Cancers Except Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study drug no longer available
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-19-19/TGen 19-001; NCI-2020-03144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0C-19-19/TGen 19-001 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — CYT003-QbG10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CMP-001, INCAGN01949) (Experimental): Patients receive CMP-001 SC on day 1 of weeks 1 and 2 and IT on day 1 of weeks 3-6 in the absence of disease progression or unacceptable toxicity. Patients also receive INCAGN01949 IT on day 1 of weeks 3-6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Agonistic Anti-OX40 Monoclonal Antibody INCAGN01949; Drug: VLP-encapsulated TLR9 Agonist CMP-001

INTERVENTIONS:
Biological: Agonistic Anti-OX40 Monoclonal Antibody INCAGN01949 — Given IT
  Other Names: Anti-OX40 Agonist Antibody INCAGN01949; Anti-OX40 Monoclonal Antibody INCAGN0194; INCAGN 1949; INCAGN-1949; INCAGN1949; Monoclonal Antibody INCAGN01949; NCAGN01949
Drug: VLP-encapsulated TLR9 Agonist CMP-001 — Given SC and IT
  Other Names: ARB-1598; CMP-001; CYT 003; CYT-003

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of CMP-001 and how well it works when given together with INCAGN01949 in treating patients with stage IV pancreatic cancer and other cancers except melanoma. CMP-001 is made up of a short piece of DNA that is packaged in a protein, known as a virus-like particle (VLP). VLPs are detected and processed by cells of the immune system. The DNA contained in CMP-001 activates the immune system and recruit cells of the immune system to the tumor. INCAGN01949 is an antibody, a type of protein, which has been shown to stimulate the immune system. Injecting CMP-001 and INCAGN01949 directly into the tumor may work against tumor cells to slow tumor growth by causing tumor cells to die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and tolerance of virus-like particle VLP-encapsulated TLR9 agonist CMP-001 (CMP-001 [TLR9 agonist]) in combination with agonistic anti-OX40 monoclonal antibody INCAGN01949 (INCAGN01949) (an activating antibody against OX40) both given intratumorally for patients with previously treated (for their metastatic disease) pancreatic ductal adenocarcinoma and other types of cancer except melanoma. (Phase IB) II. To determine the efficacy (disease control rate of complete response [CR] + partial response [PR] + stable disease [SD] X 16 weeks) of CMP001 (TLR9 agonist) in combination with INCAGN01949 (anti-OX40 antibody) for patients with previously treated (for their metastatic disease) pancreatic ductal adenocarcinoma. (Phase II) III. To determine effects on tumor markers. (Phase II)

SECONDARY OBJECTIVES:

I. Define the toxicity of the combination of CMP-001 (TLR9) + INCAGN01949 (OX40).

II. Determine progression free survival and overall survival.

EXPLORATORY OBJECTIVES:

I. Using flow cytometry on peripheral blood OX40 expression will be analyzed within the lymphocyte subsets (effector T cell [Teff] and regulatory T cell [Treg]).

II. On tissue samples collected prior to, and during, treatment, will:

IIa. Use flow cytometry to enumerate CD4+ and CD8+ T cell subsets, and the expression of activation/differentiation markers (including CD127, HLA-DR, CD45RO, CCR7, CXCR3) on each.

IIb. Use reverse transcriptase-polymerase chain reaction (RT-PCR) and sequencing to amplify and characterize the T-cell receptor (TCR)a and b sequences of tumor-infiltrating T cells, looking for evidence of oligoclonal T cell expansion, OX40 expression.

IIc. If there is adequate tumor tissue, perform ribonucleic acid sequencing (RNAseq) to determine different immune cell populations, including T cells and macrophages.

OUTLINE: This is a phase Ib, dose-escalation study of INCAGN01949, followed by a phase II study.

Patients receive CMP-001 subcutaneously (SC) on day 1 of weeks 1 and 2 and intratumorally (IT) on day 1 of weeks 3-6 in the absence of disease progression or unacceptable toxicity. Patients also receive INCAGN01949 IT on day 1 of weeks 3-6 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Histologically or cytologically confirmed pancreatic adenocarcinoma with metastasis or other locally advanced un-resectable solid tumor malignancies (during the phase Ib and pancreatic cancer during phase II) deemed appropriate by the investigator except melanoma
* Patients will have had at least 2 prior therapies for locally advanced, unresectable and/or metastatic disease. Adjuvant therapy will count as one line of therapy if disease progression occurred during treatment or within 6 months of completion. Patients with metastatic pancreatic cancer must have received either fluorouracil/Irinotecan/leucovorin calcium/oxaliplatin (FOLFIRINOX) or a gemcitabine-based regimen as one of their prior lines of therapy. Patients with germline BRCA mutations must have received olaparib as maintenance therapy
* Be willing to undergo an image-guided biopsy of a tumor lesion at baseline, after 2 weeks of IT injection and 4 weeks of IT injection (week 4 and 6), unless tumor is considered inaccessible or biopsy is otherwise considered not in the patients best interest
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Subjects must have at least one extra-central nervous system (CNS), non-bone tumor lesion amenable for IT injection >= 1.5 cm and that is not in close proximity or encasing crucial structures such as major blood vessels, trachea, nerve bundles etc. Measurable disease is required in a minimum of two lesions (one injected and one other) and there must be at least one measurable lesion in addition to the one being injected
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL without transfusions within 7 days of assessment (transfusions are allowed prior to this period)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 X ULN OR
* Aspartate transaminase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine transferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN

  * NOTE: Low molecular weight heparin at full dose or prophylactic dose is allowed as long as the treating physician deems it safe to hold the low molecular weight heparin (LMWH) on the day before and the day of the intra-tumoral injection. No other anti-coagulants are permitted
  * Because of the intratumor injections patients cannot be on any anticoagulants other than LMWH
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN

  * NOTE: Low molecular weight heparin at full dose or prophylactic dose is allowed as long as the treating physician deems it safe to hold the LMWH on the day before and the day of the intra-tumoral injection. No other anti-coagulants are permitted.
  * Because of the intratumor injections patients cannot be on any anticoagulants other than LMWH
* Female participants of childbearing potential should have a negative serum pregnancy test within 24 hours prior to receiving first dose of trial medication
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP)

    * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

      * Has not undergone a hysterectomy or bilateral oophorectomy; or
      * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 180 days after the last dose of trial treatment
* Male participants must agree to use contraception as detailed in the full protocol during the treatment period and for at least 120 days after the last dose of trial treatment and refrain from donating sperm during this period

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Investigator. If patients received prior ipilimumab or anti-CTLA4 compound and had adrenal insufficiency, treat these subjects with stress dose steroids prior to intratumoral injections. Patients may receive stress steroids orally or intravenously (IV) before the procedure
* Hypersensitivity to CMP-001 (TLR9 agonist) or INCAGN01949 (anti-OX40) or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to week 1/day 1, or who has not recovered (i.e., =< grade 1 or to baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, investigational agent, targeted small molecule therapy, or radiation therapy within 3 weeks (or 5 half-lives whichever is shorter) prior to week 1/ day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent(s)

  * Note: Patients with =< grade 2 neuropathy are an exception to this criterion and may qualify for the trial
  * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Other malignancies which have been treated with curative intent, or for which patients are not receiving active therapy, may be considered upon discussion with the investigator
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. Use of prophylactic anti-epileptic drugs is permitted. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active bacterial infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has active hepatitis B or C. Treated hepatitis C with sustained virologic response, and patients who are negative for hepatitis B surface antigen (sAg) are not excluded

  * Note: Without known history, testing needs to be performed to determine eligibility
* Current, serious, clinically significant cardiac arrhythmias as determined by the treating investigator
* Has received a live vaccine within 30 days of planned start of trial therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients must not be receiving any anticoagulation. Low molecular weight heparin at full dose or prophylactic dose is allowed as long as the treating physician deems it safe to hold the LMWH on the day before and the day of the intra-tumoral injection
* Patients should not be on aspirin or any anti-platelet agent. Patients may have been receiving aspirin 81 mg if deemed safe by the investigator to hold aspirin for the duration of the study, starting at least 7 days prior to start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Disease control rate (Phase II) | Up to 16 weeks
  Will assess complete response (CR) + partial response (PR) + stable disease (SD) via Response Evaluation Criteria in Solid Tumors (RECIST) and immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST). All proportions will be estimated using an exact 95% binomial confidence interval.
Objective response rate (CR + PR) | Up to 2 years
  Will be evaluated using the RECIST 1.1 and iRECIST. Changes (i.e. improvements) in tumor measurements from baseline values will be assigned a status of complete response (CR) or partial response (PR) or stable disease (SD). Objective response measurements will comprise the sum of CR plus PR.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  All adverse events occurring on or after week 1/day 1 will be summarized by body systems and per grade according to National Cancer Institute (NCI)-Common Terminology Criteria (CTC) version 5.
Progression free survival (PFS) | Up to 2 years
  PFS is defined as the interval from the date of registration (i.e. assignment of patient number) to the earliest date of documented evidence of recurrent or progressive disease, or the date of death due to any cause, whichever occurs first. All proportions will be estimated using an exact 95% binomial confidence interval, and a Kaplan-Meier analysis will be performed.
Overall survival | Up to 2 years
  Will be measured from the date of registration (i.e. assignment of patient number) to the date of death due to any cause, or the date of last contact (censored observations). All proportions will be estimated using an exact 95% binomial confidence interval, and a Kaplan-Meier analysis will be performed.

OTHER OUTCOMES:
OX40 expression within the lymphocyte subsets (effector T cell [Teff] and regulatory T cell [Treg]) | Up to 2 years
  Will be analyzed by flow cytometry on peripheral blood, within the lymphocyte subsets (Teffs and Tregs).
Enumeration of CD4+ and CD8+ T cell subsets | Up to 2 years
  Will be enumerated using flow cytometry.
Expression of activation/differentiation markers on CD4+ and CD8+ T cell subsets | Up to 2 years
  Will analyze CD127, HLA-DR, CD45RO, CCR7, CXCR3 using flow cytometry.
Amplification and characterization of T cell receptor (TCR) a and b sequences of tumor-infiltrating T cells | Up to 2 years
  Will be analyzed using reverse transcriptase-polymerase chain reaction (RT-PCR) and sequencing.
Immune cell populations | Up to 2 years
  Will perform ribonucleic acid sequencing (RNASeq) to determine immune cell populations including T cells and macrophages.

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Hanna, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California